CLINICAL TRIAL: NCT01334801
Title: Biomarkers in Aortic Stenosis, Hypertrophic Cardiomyopathy, Mitral Regurgitation, Aortic Regurgitation, Prosthetic Heart Valve Dysfunction, and Tricuspid Regurgitation From Pacemaker Leads Study
Brief Title: Biomarkers in Aortic Stenosis - B.A.S.S.
Acronym: BASS
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 09-006757
Record Dates: First submitted 2011-04-12; First posted 2011-04-13 (Estimated); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Aortic Stenosis; Disorder of Prosthetic Cardiac Valve; Aortic Valve Insufficiency; Mitral Valve Insufficiency; Hypertrophic Cardiomyopathy; Tricuspid Valve Insufficiency
Keywords: aortic stenosis; von Willebrand factor; mitral valve replacement; aortic valve replacement; prosthetic valve dysfunction; brain natriuretic peptide; mitral valve regurgitation; aortic valve regurgitation; hypertrophic cardiomyopathy; tricuspid insufficiency
MeSH Terms: conditions — Aortic Valve Stenosis; Aortic Valve Insufficiency; Mitral Valve Insufficiency; Cardiomyopathy, Hypertrophic; Tricuspid Valve Insufficiency | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (11):
- Aortic Stenosis: Restricted aortic valve motion and a peak Doppler aortic velocity > 2.5 m/sec blood draw
  Interventions: Procedure: Blood Draw
- Aortic regurgitation: Echocardiographic and Doppler evaluation revealing aortic regurgitation with data adequate to calculate regurgitant volume
  Interventions: Procedure: Blood Draw
- Aortic valve replacement: Mechanical or biological aortic valve replacement
  Interventions: Procedure: Blood Draw
- Mitral regurgitation: Echocardiographic and Doppler evaluation revealing mitral regurgitation with data adequate to calculate regurgitant volume
  Interventions: Procedure: Blood Draw
- Mitral valve replacement: Mechanical or biological mitral valve replacement
  Interventions: Procedure: Blood Draw
- Hypertrophic cardiomyopathy: Patients with known hypertrophic cardiomyopathy who are referred for clinically indicated echocardiography
  Interventions: Procedure: Blood Draw
- Severe TR with pacemaker / ICD lead: Patients referred for clinically indicated echocardiography who have severe tricuspid regurgitation associated with a pacemaker or defibrillator lead documented by echocardiography
  Interventions: Procedure: Blood Draw
- Prosthetic valve dysfunction: Patients with prior heart valve replacement or repair referred for clinically indicated echocardiography who demonstrate stenosis, regurgitation, dehiscence.
  Interventions: Procedure: Blood Draw
- Normal controls: Patients with no heart murmur or history of valve replacement, stenosis, regurgitation, or hypertrophic cardiomyopathy
- Left ventricular assist device patients: Patients with previously implanted LVAD
- Renal dialysis patients: Patients on hemodialysis, peritoneal dialysis, or chronic kidney disease with dialysis fistula to be created.

INTERVENTIONS:
Procedure: Blood Draw — Two tubes of blood (about five tablespoons) will be drawn for research purposes, and these will be analyzed for the following tests:
  1. BNP (Brain Natriuretic Peptide)
  2. (PFA) Platelet Function Analyzer 100
  3. von Willebrand Factor (vWF) antigen
  4. (vWF) multimers
  5. (vWF) *activity by latex aggregation
  6. Plasma stored for development of new testing approaches
  Groups: Aortic Stenosis; Aortic regurgitation; Aortic valve replacement; Hypertrophic cardiomyopathy; Mitral regurgitation; Mitral valve replacement; Prosthetic valve dysfunction; Severe TR with pacemaker / ICD lead

SUMMARY:
This study is being done to determine whether or not new blood test(s) can determine the severity of heart conditions. Aortic stenosis, hypertrophic cardiomyopathy, mitral regurgitation, aortic regurgitation, artificial heart valve regurgitation or stenosis, and tricuspid valve regurgitation associated with pacemaker leads are the cardiac disorders under study. The blood tests involve analysis for von Willebrand Factor antigen and activity, von Willebrand Factor multimers, and brain natriuretic peptide (BNP) levels. The results of the blood tests will be compared to the information from the clinically-indicated echocardiogram and one blood test compared to another.

DETAILED DESCRIPTION:
Patients with aortic stenosis, hypertrophic cardiomyopathy, mitral regurgitation, aortic regurgitation, artificial heart valve regurgitation or stenosis, and tricuspid valve regurgitation associated with pacemaker leads who are referred for clinically-indicated echocardiographic exams at Mayo Clinic, in Jacksonville, Florida will be screened for participation in the study. The plan is to have 292 people take part in this study. This minimal risk study will consist of the recording of patient data, activity and bleeding questionnaires, and collection and analysis of blood samples. Each blood sample will be analyzed for von Willebrand Factor antigen and activity, and von Willebrand Factor multimers, and BNP. Blood samples will be sent to the Mayo Special Coagulation Lab for analysis.

Objective:

This study seeks to assess the degree of association of the von Willebrand Factor activity indices and BNP to the severity of cardiac lesions, and to note a relationship between acquired bleeding the the hematologic abnormalities. Plasma will be stored in attempt to develop new in vitro tests of von Willebrand factor (VWF) activity.

ELIGIBILITY:
Inclusion Criteria:

* patients with mild, moderate, or severe aortic stenosis or aortic or mitral prosthesis. Patients with aortic or mitral regurgitation. patients with hypertrophic cardiomyopathy. Patients with dysfunctional heart valve replacement or repair. Patients with severe tricuspid regurgitation associated with pacemaker or defibrillator lead. Ten normal control patients who will not be required to have echocardiography
* referred for a clinically indicated echocardiogram; the echo must be of good quality and specifically have patient height, weight, left ventricular outflow tract diameter, subaortic velocity profile by Doppler, and aortic transvalvular continuous wave Doppler velocity profile. For mitral regurgitation and aortic regurgitation the data must be adequate to allow calculation of regurgitant volume. For hypertrophic cardiomyopathy, a recording of left ventricular outflow tract peak velocity must be recorded
* 21 years or older
* patients with aortic stenosis, defined as peak aortic velocity greater than 2.5 m/sec with evidence of aortic valve thickening, or an aortic or mitral valve prosthesis
* able to provide written informed consent

Exclusion Criteria:

* Missing or inadequate echocardiographic data
* inability to give informed consent
* inability to provide a research blood sample
* hemoglobin less than 8
* severe valvular regurgitation
* stenosis of the mitral valve

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cardiology, referred for clinically-indicated echocardiograms
Sampling Method: Non-Probability Sample
Enrollment: 378 (Actual)
Dates: Start 2010-07; Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Correlation of Von Willebrand Multimer ratio to cardiac lesion severity | 2 years
  To accomplish the specific aims, the investigators propose to collect clinical and echocardiographic data, and blood samples for von Willebrand Factor antigen and activity, von Willebrand Factor multimers, and BNP in patients with aortic stenosis, or aortic or mitral valve prosthesis, mitral regurgitation, hypertrophic cardiomyopathy, aortic regurgitation, and tricuspid regurgitation associated with pacemaker or defibrillator.

SECONDARY OUTCOMES:
Correlation of other VWF activity measures with cardiac lesion severity. | 2 years
  Comprehensively analyze the ability of VWF indices to discriminate severe from non-severe valvular disease, prosthetic valve dysfunction, and describe the prevalence of VWF abnormalities in this wide range of cardiac lesions associated with intravascular turbulence.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph L Blackshear, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Jacksonville, Florida, United States

REFERENCES:
- [Derived] Blackshear JL, Stark ME, Agnew RC, Moussa ID, Safford RE, Shapiro BP, Waldo OA, Chen D. Remission of recurrent gastrointestinal bleeding after septal reduction therapy in patients with hypertrophic obstructive cardiomyopathy-associated acquired von Willebrand syndrome. J Thromb Haemost. 2015 Feb;13(2):191-6. doi: 10.1111/jth.12780. Epub 2014 Dec 12. PMID 25387993
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials